CLINICAL TRIAL: NCT06786117
Title: Swallowing in Obstructive Sleep Apnea (OSA) & Continuous Positive Airway Pressure (CPAP) Intolerance
Brief Title: Swallowing in OSA & CPAP Intolerance
Acronym: SLP-PAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Denise Dewald (Other)
Collaborators: American Academy of Sleep Medicine (Other); Case Western Reserve University (Other); MetroHealth Medical Center (Other)
Responsible Party: Sponsor-Investigator, Denise Dewald, Faculty, Pulmonary, Critical Care and Sleep Medicine- Department of Medicine, MetroHealth Medical Center
Organization: MetroHealth Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY0000450; 299-JF-23 (Other Grant/Funding Number: American Academy of Sleep Medicine (AASM) Foundation)
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea, Obstructive; Healthy
Keywords: OSA; obstructive sleep apnea; sleep apnea; myofunctional therapy; swallowing exercises; speech language pathology; modified barium swallow; CPAP; CPAP intolerance; CPAP adherence; continuous positive airway pressure; EMST-150; expiratory muscle strength training; respiratory muscle strength; respiratory muscle strength training; non-snorers
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Myofunctional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healthy airways group (No Intervention): Participants will get a home sleep test to verify that sleep disordered breathing is not present. They will do a modified barium study (MBS) and a measurement visit to assess oral and respiratory muscle strength, nasal airflow, tongue mobility, eating and drinking, dental and facial form, and posture. They will also fill out some questionnaires.
- Successful CPAP user (No Intervention): Participants who do well will CPAP will do a modified barium study (MBS) and a measurement visit to assess oral and respiratory muscle strength, tongue mobility, nasal airflow, eating and drinking, dental and facial form, and posture. They will also fill out some questionnaires. Participants will also provide their CPAP data on an SD card. Participants will also do a home sleep test if there is no recent sleep study available.
- CPAP intolerant - SLP exercises only (Experimental): CPAP intolerant participants will try to use CPAP for two weeks with individualized coaching. If they still have problems with CPAP, they will do a modified barium study (MBS), a baseline home sleep test, and a measurement visit. During the measurement visit their oral and respiratory strength, nasal airflow, tongue mobility, eating and drinking, dental and facial form, and posture will be assessed. They will also fill out questionnaires.
  Participants with abnormalities on their MBS will get a 7-week course of standard swallowing exercises, with weekly in-person visits with a speech pathologist. They will be expected to do daily exercises (which will take 20-30 minutes). They will then try to use CPAP for two weeks to see if they are able to use CPAP better.
  If they do well with CPAP or are still struggling with CPAP but do not want to continue onto the myofunctional therapy arm, they will do an MBS, home sleep test, questionnaires, and the measurement visit again.
  Interventions: Other: SLP swallowing exercises
- CPAP intolerant - OMT exercises only (Experimental): CPAP intolerant participants will try to use CPAP for two weeks with individualized coaching. If they still have problems with CPAP, they will do a modified barium study (MBS), a baseline home sleep test, and also a measurement visit. During the measurement visit their oral and respiratory strength, tongue mobility, nasal airflow, eating and drinking, dental and facial form, and posture will be assessed. They will also fill out some questionnaires.
  CPAP intolerant participants without abnormalities on their MBS will get oral myofunctional therapy (OMT) exercises. The course of exercises will take 7 weeks to complete, with weekly video follow up visits. The exercises will take 20-30 minutes to do over the course of the day.
  After completing the 7-week course, participants will repeat the home sleep test, modified barium study, questionnaires, and measurement visit, and will once more try using CPAP for two weeks to see if they are able to use CPAP better.
  Interventions: Other: myofunctional exercises
- CPAP intolerant - SLP and OMT (Experimental): CPAP intolerant participants will try to use CPAP for two weeks with individualized coaching. If they still have problems with CPAP, they will do a modified barium study (MBS), a baseline home sleep test, and also a measurement visit. During the measurement visit their oral and respiratory strength, nasal airflow, tongue mobility, eating and drinking, dental and facial form, and posture will be assessed. They will also fill out questionnaires.
  Participants with abnormalities on their MBS will get standard swallowing exercises based on the abnormalities. They will then try using CPAP for two weeks. If they do not improve their CPAP tolerance with standard swallowing exercises, they will do a course of myofunctional therapy exercises. Both courses will be 7 weeks long, with daily exercises to do at home lasting 20-30 min.
  They will then repeat the home sleep test, MBS, questionnaires, and measurement visit, and will try using CPAP for two weeks to see if they can use CPAP better.
  Interventions: Other: SLP swallowing exercises; Other: myofunctional exercises

INTERVENTIONS:
Other: SLP swallowing exercises — Clinical speech language pathologists will provide standard exercises based on the abnormalities seen on the modified barium swallow. Exercises are expected to include the effortful swallow, the Mendelsohn maneuver, expiratory muscle strength training with the EMST-150, supraglottic swallow, super supraglottic swallow, chin tuck against resistance isokinetic exercise, chin tuck against resistance isometric exercise, Masako maneuver, Shaker isometric head lift exercise, Shaker isokinetic head lift exercise, Falsetto high pitch glide exercise, tongue press exercise
  Other Names: speech language pathology exercises; SLP exercises
  Arms: CPAP intolerant - SLP and OMT; CPAP intolerant - SLP exercises only
Other: myofunctional exercises — Participants will get a variety of exercises aimed at improving bolus formation, strengthening the seal of the soft palate with the tongue, and habituating nasal breathing. There will also be exercises aimed at stabilizing the epiglottis and strengthening the muscles supporting the lateral pharyngeal walls. Expiratory muscle strength training with the EMST-150 will also be done.
  Other Names: orofacial myofunctional therapy (OMT); OMT exercises
  Arms: CPAP intolerant - OMT exercises only; CPAP intolerant - SLP and OMT

SUMMARY:
This study has two parts: an observational part and an interventional part.

The goal of the observational part of the study is to look for variations in swallowing in adults with obstructive sleep apnea (OSA) and in adults who don't snore. The main questions it aims to answer are:

* Are there differences in swallowing between people with OSA and people who don't snore?
* Are there differences in swallowing between people with OSA who do well with continuous positive airway pressure (CPAP) therapy and those who struggle with CPAP?

This may help us better understand what causes OSA, which may help us develop alternate ways to treat or even prevent OSA. It may also help us improve care for people with OSA who struggle with CPAP. Participants will be aged 40-60 years, except women up to the age of 70 will be included in the healthy control (non-snorer) group.

Participants will:

* Undergo a type of x-ray study called a modified barium swallow study (MBS)
* Come to MetroHealth Medical Center for a measurement visit to:

  * assess the strength of their tongue, lips, and cheeks
  * assess the strength of their breathing muscles
  * assess for restrictions in tongue mobility (tongue ties)
  * observe their resting breathing
  * take photos of their mouth and posture
  * take videos of them drinking and eating
* Complete some questionnaires
* For successful CPAP users: we will download data from the chip in their CPAP device
* Do a home sleep test (except for successful CPAP users who have had a recent in-lab sleep test)

The goal of the interventional part of the study is to test swallowing exercises in people ages 40-60 years with OSA who struggle with CPAP. The main question it aims to answer is:

• Can swallowing exercises help people who struggle with CPAP sleep better with CPAP?

Participants will:

* Try to use CPAP for 2 weeks with individualized support
* Do all the investigations listed in the observational part of the study
* Do one or two courses of swallowing exercises, each of which would last 7 weeks. Participants will be asked to do daily exercises; exercises will take 20-30 minutes to perform.
* Try to use CPAP for 2 weeks after the course of exercises
* Repeat the investigations listed in the observational part of the study to see if changes occurred with the swallowing exercise intervention.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder in which the throat narrows abnormally or even collapses fully during sleep. The narrowing leads to sleep disruption and increases the risk of many chronic health conditions. We do not understand why the throat narrows in some people during sleep but not in others. While being overweight or obese increases a person's risk of OSA, it is only one part of the problem. Some thin adults and children have OSA, and many overweight or obese people do not have OSA. In addition, many people with OSA struggle to benefit from current OSA treatments like continuous positive airway pressure (CPAP), which uses air pressure to hold the airway open during sleep. We need improved understanding of OSA in order to improve treatment of it.

The throat is used for swallowing as well as for breathing. Hence it should not be surprising if a throat that has trouble staying open during sleep might also have some abnormalities during swallowing. Indeed, some research has shown subtle abnormalities in swallowing in people who have snoring or OSA compared to people who don't snore at all. We would like to further develop this line of research.

This study has two arms: an observational arm to look for differences in swallowing, and an interventional arm to see if swallowing exercises can improve people's ability to use CPAP.

The purpose of the observational arm is to look for differences in swallowing between healthy people and people who have obstructive sleep apnea (OSA) using a variety of measurement techniques, some of which have not been done in the past. Understanding the differences in swallowing may help us to develop new treatments for OSA. It may also help us to figure out how to prevent OSA from developing in the first place. We are also looking to see if there are swallowing differences between people with OSA who don't tolerate CPAP compared to people who do well with CPAP. If there are differences, these differences may help us better understand why some people do not tolerate CPAP, and may lead to the development of novel treatments such as exercise therapies to help them do better with CPAP.

The interventional arm will test exercise therapies to see if they will help people who struggle with CPAP. The goal is not to cure OSA, but to help people be able to use CPAP better so that they can sleep better. Participants who have abnormalities in their swallowing study will get exercises from speech language pathologists (SLP, also known as speech therapists) aimed at trying to correct those abnormalities. Participants will then try to use CPAP again. Participants who still can't sleep well with CPAP after those exercises, or who don't have abnormalities on the swallowing study, will get another type of exercise therapy based on an exercise technique called orofacial myofunctional therapy (OMT). This therapy aims to train exclusive nasal breathing and correct variations in the swallow. This sort of exercise technique has had some success in improving CPAP use as well as in reducing the severity of OSA. We have created a streamlined exercise protocol based on these techniques that we hope will provide better results in a shorter period of time. At the end of the exercise interventions, the participants will repeat the investigations that were done at the beginning of the study.

Investigations will include home sleep testing, CPAP trials (only for participants with OSA and CPAP intolerance), a modified barium swallow study (MBS), a measurement visit, and questionnaires. During the measurement visit, there will be assessments of the strength of the tongue, lips, and cheeks, assessment of nasal airflow, respiratory muscle strength, restrictions in tongue mobility (tongue tie), posture, dental and facial form, and eating and drinking. The modified barium swallow study uses x-rays; the amount of radiation from the procedure is about what a person would receive from about 4.5 months of background radiation. It is a little bit more radiation than what a person would receive from a mammogram, but much less than what a person would receive from a CT scan.

ELIGIBILITY:
Inclusion Criteria for healthy airways participants:

* Naturally ideal dental occlusion without orthodontic intervention, including successful eruption of wisdom teeth (without significant dental crowding, though minor rotation of less than 4 teeth will be acceptable)
* No sleep-related complaints
* No snoring.
* They should be missing no more than 4 of their natural teeth, and these should have been lost to decay or accident rather than due to crowding. A person whose wisdom teeth came in successfully but were extracted "preventatively" will be eligible for the study.
* Should be getting at least 6 hours of sleep nightly.
* BMI between 18.5 and 35

Inclusion Criteria for participants with OSA who are successful CPAP users:

* Participant will have experienced significant benefits from therapy and have had such benefit since the first night of use. Participant should have no significant sleep complaints when using CPAP.
* Uses CPAP > 6 hours of nightly use on > 90% of nights using a nasal mask.
* Residual device AHI < 5 events/hour.
* Has used CPAP for at least 12 months.
* Symptomatic at diagnosis, with polysomnography (PSG) showing AASM AHI 5-60 and symptoms attributable to OSA, with greater than 75% of the apneas and hypopneas being obstructive in nature. Home sleep apnea testing (HSAT) will also be accepted, with RDI 5-60, with greater than 75% of the apneas and hypopneas being obstructive in nature.
* Should be getting at least 6 hours of sleep nightly.
* BMI between 18.5 and 35

Inclusion Criteria for participants with OSA who have CPAP intolerance:

* Symptomatic, with polysomnography (PSG) showing AASM AHI 5-60 and symptoms attributable to OSA, with greater than 75% of the apneas and hypopneas being obstructive in nature. Home sleep apnea testing (HSAT) will also be accepted, with RDI 5-60, with greater than 75% of the apneas and hypopneas being obstructive in nature.
* Attempted nightly use for at least 2 weeks (at least 12/14 nights), with average use < 4 hours, and difficulty tolerating PAP during a titration study, with complaints of difficulty breathing with CPAP or other difficulties that are not clearly related to identifiable causes (claustrophobia, mask discomfort, untreated RLS, untreated mouth leak, poor sleep hygiene, drug use, etc.).
* Must be able to breathe through their noses comfortably while awake.
* Able and willing to do daily swallowing exercises (15-30 minutes per day) for a total of 14 weeks.
* Able and willing to use a positional therapy device to avoid supine sleep and to adjust their CPAP device settings (instructions will be provided).
* BMI between 18.5 and 35
* Not actively undergoing bariatric treatment or planning to start bariatric treatment within the next 6 months.

Exclusion Criteria for all participants:

* Presence of symptomatic swallowing disorders, neuromuscular disorders affecting the upper airway, or neurodegenerative disorders.
* Co-existing sleep disorders such as narcolepsy, untreated restless legs syndrome, circadian rhythm disorders, or behavioral insomnia/poor sleep hygiene.
* Clinically significant congenital or acquired anomalies or history of surgery on the head and neck, excluding adenotonsillectomy, turbinate reduction, and septoplasty. Participants who had a tongue tie release outside of the newborn period will be excluded, but those who had tongue tie release in the newborn period will be eligible.
* Known complex sleep apnea or a history of conditions that are associated with the development of complex sleep apnea, such as heart failure, atrial fibrillation, a history of stroke, or opioid use.
* Prescription or nonprescription stimulant use (excluding caffeine).
* Substance use disorder or nightly alcohol consumption, as these significantly interfere with normal sleep.
* Current unstable illness (such as asthma, hypertension, cancer, etc.), kidney failure with restrictions on fluid consumption, or unplanned hospitalization in the past year for an ongoing condition.
* Risk factors for harm from expiratory strength testing and training: history of spontaneous pneumothorax, presence of CSF drain, recent trauma involving head, neck, or chest, history of recurrent epistaxis, history of esophageal surgery, active or recent hemoptysis, history of lung transplant or lung resection, eardrum rupture or any other condition of the ear, uncontrolled gastroesophageal reflux, abdominal hernia or recent hernia repair, urinary or fecal incontinence, presence of aneurysm (such as cerebral or aortic).
* Participants with CPAP intolerance only: Latex allergy in themselves or household members (due to balloon use in exercises).
* Allergy to Micropore paper tape (used in home sleep testing and for participants with CPAP intolerance during 2-week CPAP trial and exercise intervention).
* Pregnancy, actively trying to get pregnant, or sexually active and not using birth control (for people of child-bearing potential).
* Has a condition that increases the risk of developing cancer, such as BRCA1/2.
* Does not speak English fluently.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of premature spillage in participants with OSA who are CPAP intolerant vs participants who are successful nasal CPAP users or who have healthy airways | at the time of MBS (within 2-4 weeks of study enrollment)
  MBS images will be evaluated for premature spillage during oral bolus formation. Comparison of prevalence of premature spillage will be made between study groups.
Effect of swallowing exercise intervention for CPAP intolerance | 3-7 months after enrollment
  The effect of a swallowing exercise intervention on CPAP intolerance will be assessed, as reflected by change in usage from the participants' own pre-treatment CPAP data.
  The results of the two exercise interventions will be pooled, as the goal is to see if swallowing exercises can improve CPAP tolerance rather than to compare therapies.

SECONDARY OUTCOMES:
Baseline length of the oropharyngeal seal during bolus formation in the modified barium swallow study (MBS) | at the time of MBS (within 2-4 weeks of study enrollment)
  The length of the oropharyngeal seal during bolus formation will be measured to assess for differences between participants with healthy airways and those with OSA.
Baseline breathing route during wakefulness as assessed by MBS | at the time of MBS (within 2-4 weeks of study enrollment)
  Breathing route (oral, oronasal, or nasal) will be determined by soft palate position during resting breathing under fluoroscopy in the modified barium swallow study. Comparison will be made between healthy airways, CPAP intolerant, and successful CPAP user groups.
Baseline tongue position as observed during nasal breathing during MBS | at the time of MBS (within 2-4 weeks of study enrollment)
  A high or low tongue resting position during nasal breathing will be noted upon review of the MBS images. Tongue position will be compared between study groups.
Baseline soft palate shape as observed during nasal breathing during MBS | at the time of MBS (within 2-4 weeks of study enrollment)
  Assessment of the angulation of the soft palate during nasal breathing will be performed. Results will be compared between healthy airways, CPAP intolerant, and successful CPAP user groups.
Baseline assessment of Tipper- vs Dipper-type oral swallowing | at the time of MBS (within 2-4 weeks of study enrollment)
  The presence of Tipper-type vs Dipper-type oral swallowing will be assessed by MBS. The prevalence of the oral swallowing types in the study groups will be compared.
Baseline assessment of anterior tongue strength | at the time of the measurement visit (within 2-4 weeks of study enrollment); participants with CPAP intolerance will have a second measurement visit at the end of the study
  Assessment of anterior tongue strength will be made using an IOPI (Iowa Oral Performance Index) system. Strength will be compared between groups.
Baseline assessment of posterior tongue strength | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Assessment of posterior tongue strength will be made using an IOPI (Iowa Oral Performance Index) system. Strength will be compared between groups.
Baseline assessment of combined lip/cheek strength | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Assessment of combined lip/cheek strength will be made using an IOPI (Iowa Oral Performance Index) system. Strength will be compared between groups.
Baseline assessment of combined lip/cheek activation during swallowing | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Assessment of combined lip/cheek activation during swallowing will be made using an IOPI (Iowa Oral Performance Index) system. Extent of combined lip/cheek activation during swallowing will be compared between groups.
Baseline maximum expiratory pressure | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Maximum expiratory pressure (MEP) will be assessed and compared between study groups.
Baseline maximum inspiratory pressure via oral route | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Maximum inspiratory pressure by the oral route will be assessed and compared between study groups.
Baseline sniff inspiratory pressure (SNIP) via nasal route | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Baseline maximum sniff inspiratory pressure (SNIP) by the nasal route will be assessed and compared between study groups.
Baseline awake resting breathing route assessment by nasal pressure signal | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Awake breathing route (oral, oronasal, or nasal) will be inferred by nasal pressure signal during resting breathing. Comparison will be made between healthy airways, CPAP intolerant, and successful CPAP user groups.
Baseline assessment of Mallampati score | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Mallampati score will be assessed by physical examination. Comparisons will be made between study groups.
Baseline assessment of Friedman tongue position score | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Friedman tongue position score will be assessed by physical examination. Comparisons will be made between study groups.
Baseline anterior tongue tie evaluation | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Anterior tongue tie evaluation will be made using the tongue tie assessment tool. Comparisons between groups will be made.
Baseline posterior tongue tie evaluation | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Posterior tongue tie evaluation will be made using the tongue tie assessment tool. Comparisons between groups will be made.
Baseline visual differences in swallowing | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Utilization of lip and cheek muscles during swallowing will be assessed visually (with videorecording). Comparisons will be made between the study groups.
Baseline head tilt angle differences | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Head tilt angle will be measured by glasses with an attached digital level. Comparisons will be made between study groups.
Baseline postural assessment | at the time of the measurement visit (within 2-4 weeks of study enrollment)
  Photographs will be taken with the participant standing next to a plumb line for postural assessment. Comparisons will be made between study groups.
Baseline CPAP waveform differences between participants with CPAP intolerance and participants who are successful CPAP users (participants with OSA only) | At study enrollment (successful CPAP users) or after baseline 2-week CPAP trial (participants with CPAP intolerance), within 1 months of enrollment
  CPAP waveforms will be assessed for the presence of negative effort dependence or other differences in the airflow waveform shapes in participants with CPAP intolerance compared to participants who are successful nasal CPAP users.
Baseline differences in nasal pressure signal during sleep between participants with CPAP intolerance and participants who are successful CPAP users (participants with OSA only) | At enrollment (if recent PSG is already available) or after completion of home sleep testing, within one month of enrollment
  Nasal pressure waveforms during sleep will be assessed for the presence of negative effort dependence or other features that may be different between participants with CPAP intolerance compared to participants who are successful nasal CPAP users, as seen in polysomnography or home sleep testing.
Baseline Swallowing Disturbance Questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Swallowing Disturbance Questionnaire. Responses will be compared between study groups.
Baseline Epworth Sleepiness Scale (ESS) | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Epworth Sleepiness Scale (ESS) questionnaire. Comparisons will be made between study groups.
Baseline Pittsburgh Sleep Quality Index (PSQI) questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Comparisons will be made between study groups.
Baseline Insomnia Severity Index (ISI) questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Insomnia Severity Index (ISI) questionnaire. Comparisons will be made between study groups.
Baseline Short Calgary Sleep Apnea Quality Of Life Index questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Short Calgary Sleep Apnea Quality Of Life Index questionnaire. Comparisons will be made between study groups.
Baseline Short Form Health Survey-36 questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the Short Form Health Survey-36 questionnaire. Comparisons will be made between study groups.
Baseline PROMIS Sleep Disturbance short form 8b questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the PROMIS Sleep Disturbance short form 8b questionnaire. Comparisons will be made between study groups.
Baseline PROMIS Sleep-related impairment short form 8a questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete the PROMIS Sleep-related impairment short form 8a questionnaire. Comparisons will be made between study groups.
Baseline sleep habits and swallowing and CPAP observations questionnaire | When baseline questionnaires are returned, within one month of enrollment.
  Participants will complete questionnaires on sleep habits and swallowing and CPAP observations. Responses will be compared between study groups.
Post-intervention assessment of AHI by home sleep testing (participants with CPAP intolerance only) | Before the post-intervention CPAP trial or two weeks after the CPAP trial, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Repeat home sleep testing will be performed after the final swallowing exercise intervention has been completed (before the CPAP trial or two weeks after the CPAP trial). Results will be compared with the participant's baseline home sleep test.
Post-intervention changes in nasal airflow during sleep (participants with CPAP intolerance only) | Before the post-intervention CPAP trial or two weeks after the CPAP trial, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Nasal pressure signal on home sleep testing will be assessed for changes in flow limitation and negative effort dependence after the intervention, and compared to the participant's pre-intervention waveforms.
Post-intervention assessment of pulse oxygen nadir by home sleep testing (participants with CPAP intolerance only) | Before the post-intervention CPAP trial or two weeks after the CPAP trial, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Repeat home sleep testing will be performed after the final swallowing exercise intervention has been completed (before the CPAP trial or two weeks after the CPAP trial). Pulse oxygen nadir will be determined and compared with the participant's baseline home sleep test.
Post-intervention assessment of time with oxygen saturation less than 90% during home sleep testing (participants with CPAP intolerance only) | Before the post-intervention CPAP trial or two weeks after the CPAP trial, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Repeat home sleep testing will be performed after the final swallowing exercise intervention has been completed (before the CPAP trial or two weeks after the CPAP trial). The time spent with oxygen saturation less than 90% will be determined and compared with the participant's baseline home sleep study.
Post-intervention differences in nasal pressure signal during home sleep testing (participants with CPAP intolerance only) | After the post-intervention 2-week CPAP trial, 3-7 months after study enrollment
  Post-intervention nasal pressure waveforms during home sleep testing will be assessed for the presence of negative effort dependence or other changes. Results will be compared to participant's baseline results and to those of participants who are successful nasal CPAP users, as seen in polysomnography or home sleep testing.
Post-intervention assessment of oral bolus formation during MBS (participants with CPAP intolerance only) | Within 2-4 weeks of the completion of the final swallowing exercise intervention, which will be 3-7 months after enrollment
  Repeat MBS after the swallowing exercise intervention will be done to assess for any changes in oral bolus formation/premature spillage.
Post-intervention length of oropharyngeal seal during bolus formation in modified barium swallow study (MBS) (participants with CPAP intolerance only) | at the time of the post-intervention MBS, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  The length of the oropharyngeal seal during oral bolus formation will be measured on MBS. Results will be compared to the participant's baseline MBS.
Post-intervention breathing route during wakefulness by MBS (participants with CPAP intolerance only) | at the time of the post-intervention MBS, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Breathing route (oral, oronasal, or nasal) will be determined by soft palate position during resting breathing under fluoroscopy in the repeat modified barium swallow study, to be done after completion of the final exercise intervention. Comparison will be made to the participant's baseline results.
Post-intervention tongue position as observed during nasal breathing during MBS (participants with CPAP intolerance only) | at the time of the post-intervention MBS, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  A high or low tongue resting position during nasal breathing will be noted upon review of the MBS images. Tongue position will be compared to participant's baseline results.
Post-intervention soft palate shape as observed during nasal breathing during MBS (participants with CPAP intolerance only) | at time of the post-intervention MBS, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Assessment of the angulation of the soft palate during nasal breathing will be performed. Results will be compared to the participant's baseline.
Post-intervention assessment of Tipper- vs Dipper-type swallowing (participants with CPAP intolerance only) | at the time of the post-intervention MBS, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  The presence of Tipper-type vs Dipper-type oral swallowing will be assessed by repeat MBS. The results will be compared to the participant's baseline.
Post-intervention assessment of anterior tongue strength (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Assessment of anterior tongue strength will be made using an IOPI (Iowa Oral Performance Index) system during the post-intervention measurement visit. Strength will be compared to participant's baseline and to baseline results for the other study groups.
Post-intervention assessment of posterior tongue strength (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Assessment of posterior tongue strength will be made using an IOPI (Iowa Oral Performance Index) system during the post-intervention measurement visit. Strength will be compared to participant's baseline and to baseline results for the other study groups.
Post-intervention assessment of combined lip/cheek strength (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Assessment of combined lip/cheek strength will be made using an IOPI (Iowa Oral Performance Index) system during the post-intervention measurement visit. Strength will be compared to participant's baseline and to baseline results for the other study groups.
Post-intervention assessment of combined lip/cheek activation during swallowing (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Repeat assessment of combined lip/cheek activation during swallowing will be made using an IOPI (Iowa Oral Performance Index) system. Extent of lip/cheek activation during swallowing will be compared to participant's baseline results and also to the baseline results of the other study groups.
Post-intervention maximum expiratory pressure (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Maximum expiratory pressure (MEP) will be assessed post-intervention and compared to participant's baseline and the baseline results of the other study groups.
Post-intervention maximum inspiratory pressure via oral route (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Maximum inspiratory pressure by the oral route will be assessed post-intervention. Results will be compared to participant's baseline results and to baseline results of other study groups.
Post-intervention sniff inspiratory pressure (SNIP) via nasal route (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention maximum sniff inspiratory pressure (SNIP) by the nasal route will be assessed. Results will be compared to participant's baseline values and between those of the other study groups.
Post-intervention awake resting breathing route assessment by nasal pressure signal (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention awake breathing route (oral, oronasal, or nasal) will be determined by nasal pressure signal during resting breathing. Comparison will be made to participant's baseline results and to those of the other study groups.
Post-intervention assessment of Mallampati score (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention Mallampati score will be assessed by physical examination. Comparisons will be made to participant's baseline value and to the Mallampati scores of the other study groups.
Post-intervention assessment of Friedman tongue position score (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention Friedman tongue position score will be assessed by physical examination. Comparisons will be made to participant's baseline score and also to scores of the other study groups.
Post-intervention anterior tongue tie evaluation (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Repeat anterior tongue tie evaluation will be made using the tongue tie assessment tool. Comparisons to participant's baseline results and the results of other study groups will be made.
Post-intervention posterior tongue tie evaluation (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention posterior tongue tie evaluation will be made using the tongue tie assessment tool. Result will be compared to participant's baseline result and to the results of the other study groups.
Post-intervention visual differences in swallowing (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention utilization of lip and cheek muscles during swallowing will be assessed visually (with videorecording). Comparisons will be made to the participant's baseline results and to the results of the other study groups.
Post-intervention head tilt angle differences (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention head tilt angle will be measured by glasses with an attached digital level. Comparisons will be made to participant's baseline value and to those of the other study groups.
Post-intervention postural assessment (participants with CPAP intolerance only) | at the time of the post-intervention measurement visit, approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Post-intervention photographs will be taken with the participant standing next to a plumb line for postural assessment. Comparisons will be made to participant's baseline results and to those of the other study groups.
Post-intervention CPAP waveform differences (participants with CPAP intolerance only) | After the post-intervention 2-week CPAP trial, 3-7 months after study enrollment.
  After the final 2-week CPAP trial, CPAP waveforms will be obtained from the CPAP data chip and assessed for the presence of negative effort dependence or other differences in the airflow waveform shapes. Results will be compared to participant's pre-intervention results and those of participants who are successful nasal CPAP users.
Post-intervention CPAP residual AHI (participants with CPAP intolerance only) | After the post-intervention 2-week CPAP trial, 3-7 months after study enrollment.
  Residual AHI will be collected from the CPAP data chip after 2-week CPAP trial at the end of the swallowing exercise intervention. Results will be compared to participant's pre-intervention results and those of participants who are successful nasal CPAP users.
Post-intervention number of nightly CPAP mask removals (participants with CPAP intolerance only) | After the post-intervention 2-week CPAP trial, 3-7 months after study enrollment.
  The number of nightly CPAP mask removals will be collected from the CPAP data chip after 2-week CPAP trial at the end of the swallowing exercise intervention. Results will be compared to participant's pre-intervention results and those of participants who are successful nasal CPAP users.
Post-intervention Swallowing Disturbance Questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second Swallowing Disturbance Questionnaire after completing the final exercise intervention. Responses will be compared to their baseline questionnaire.
Post-intervention Epworth Sleepiness Scale (ESS) (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second Epworth Sleepiness Scale (ESS) questionnaire after completing the final exercise intervention. Comparison will be made to the participant's baseline results.
Post-intervention Pittsburgh Sleep Quality Index (PSQI) questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second Pittsburgh Sleep Quality Index (PSQI) questionnaire after completing the final exercise intervention. Comparison will be made to participant's baseline results.
Post-intervention Insomnia Severity Index (ISI) questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second Insomnia Severity Index (ISI) questionnaire after completing the final exercise intervention. Comparison will be made to participant's baseline results.
Post-intervention Short Calgary Sleep Apnea Quality Of Life Index questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second Short Calgary Sleep Apnea Quality Of Life Index questionnaire after completing the final exercise intervention. Comparison will be made to participant's baseline results.
Post-intervention Short Form Health Survey-36 questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants with CPAP intolerance will complete a second Short Form Health Survey-36 questionnaire after completion of the exercise intervention(s). Comparisons will be made to their responses on the baseline questionnaire.
Post-intervention PROMIS Sleep Disturbance short form 8b questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second PROMIS Sleep Disturbance short form 8b questionnaire after completing the final exercise intervention. Comparison will be made to participant's baseline results.
Post-intervention PROMIS Sleep-related impairment short form 8a questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete a second PROMIS Sleep-related impairment short form 8a after completing the final exercise intervention. Comparison will be made to participant's baseline results.
Post-intervention sleep habits and swallowing and CPAP observations questionnaire (participants with CPAP intolerance only) | When the post-intervention questionnaires are returned, which will be approximately 3-7 months after enrollment, depending on whether one or two courses of exercises is done
  Participants will complete repeat questionnaires on sleep habits and swallowing and CPAP observations after completing the final exercise intervention. Comparison will be made to participant's baseline results.

OTHER OUTCOMES:
Long term outcome of swallowing exercise intervention on average nightly hours of CPAP use (participants with CPAP intolerance only) | 3-15 months after completion of the final exercise intervention (depending on whether participant will need a CPAP device)
  Assess long-term impact of goal-oriented oromuscular rehabilitation in OSA participants with CPAP intolerance by following up on average nightly hours of CPAP use with CPAP compliance downloads and phone follow-up, to be done 3, 6, and 12 months after the end of the final CPAP trial.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Dewald, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IDP collected throughout the trial.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning year 1 after first publication with no end date.
Access Criteria: No data use agreement or data request will be required.